CLINICAL TRIAL: NCT03260036
Title: The Effect of Bariatric Surgery on Hepatic Urea Nitrogen Handling and Cognitive Functions in Patients With Severe Non-alcoholic Fatty Liver Disease
Brief Title: Hepatic Urea Nitrogen Handling in Patients With NASH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: FHNC-bariatric
Record Dates: First submitted 2017-08-16; First posted 2017-08-24 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Urea synthesis; Ammonia; Bariatric surgery
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver tissue Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the project is to investigate the metabolic regulation of the hepatic urea nitrogen handling and various cognitive functions measured by psychometric and neurophysiological tests before and after bariatric surgery in patients with non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
NAFLD is the most common cause of chronic liver disease in the western world affecting 10-30% of the general population. It is strongly associated with the metabolic syndrome caused by overweight and obesity. NAFLD is a spectrum of liver disease ranging from steatosis (hepatocytic fat accumulation occurs without hepatocellular injury), to non-alcoholic steatohepatitis (NASH) (steatosis is accompanied by inflammation and hepatocyte injury with or without fibrosis) and to cirrhosis in patients that are not consuming excessive alcohol. The prognosis of patients with simple steatosis appears benign whereas NASH often has a progressive course with increased liver-related morbidity and mortality.

Patients with liver disease often have impairment of metabolic liver functions. The liver has numerous functions, which are essential for maintenance of life e.g. urea synthesis. This function is central in whole body nitrogen (N) homeostasis and removes ammonia, which is produced during N conversion and is extremely toxic especially for brain functions. Impairment of urea synthesis causes increased ammonia concentrations in the blood, which is taken up by the brain and contributes to development of hepatic encephalopathy in patients with liver disease. This condition is one of the most debilitating complications of liver disease as it affects cognitive functions and with increasing severity also behaviour and motor function. The mild stage (termed minimal hepatic encephalopathy) causes subtle cognitive dysfunction, which can only be detected by means of special tests. The more severe stages (manifest hepatic encephalopathy) are accompanied by manifest dysfunction of sleep pattern and orientation eventually leading to liver coma. The condition is reversible and no structural brain damage occurs.

We seek to investigate the consequences of bariatric surgery on liver and brain function with a special focus on NASH patients. The investigations will comprise examination of the capacity for urea synthesis and various psychometric and neurophysiological tests to evaluate the patient's cognitive functions before and 18 months after surgery.

A liver biopsy will be availed at the time of surgical intervention and genetic and functional characterization of urea cycle enzymes will be performed to correlate with histological scores, clinical disease staging and ammonia/capacity for urea synthesis. A further liver biopsy will be performed after 18 months to determine if there has been any change in NAFLD disease stage and urea cycle enzymes after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Referred for bariatric surgery (BMI > 40 kg/m2 or BMI > 35 kg/m2 and obesity-related complications
* Steatosis on ultrasound (US)
* Alcohol intake < 40g/day
* Exclusion of other liver diseases

Exclusion Criteria:

* Chronic inflammatory diseases
* Acute severe bacterial infection (sepsis, pneumonia, urinary tract infection etc.)
* Cancer
* Neurological diseases
* Prednisolone treatment within the last 8 weeks
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients referred for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-08-21 (Estimated)

PRIMARY OUTCOMES:
Changes in Functional Hepatic Nitrogen Clearance (FHNC) | Baseline and 18 months
  FHNC is a validated method for assessing the conversion of amino-nitrogen to urea-nitrogen by the liver

SECONDARY OUTCOMES:
Urea cycle enzymes (protein and gene level) | Baseline and 18 months
  Examined in liver biopsy
Changes in The Portosystemic Encephalopathy Syndrome-Test | Baseline and 18 months
  To evaluate changes in the patient's cognitive functions
Changes in Continuous Reaction Time Test | Baseline and 18 months
  To evaluate changes in the patient's cognitive functions
Changes in Critical Flicker Frequency | Baseline and 18 months
  To evaluate changes in the patient's cognitive functions
Changes in EEG | Baseline and 18 months
  To evaluate potential changes in the patient's EEG

CONTACTS AND LOCATIONS:
Overall Officials: Karen Louise Thomsen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No